CLINICAL TRIAL: NCT04976933
Title: Design and Feasibility of mHealth App for Pediatric Medication Adherence Post-discharge for Hematopoietic Stem Cell Transplant
Brief Title: Post-HSCT Medication Adherence mHealth App
Status: Completed | Type: Observational
Sponsor: Micah Skeens (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Sponsor-Investigator, Micah Skeens, Nurse Scientist/Principal Investigator, Nationwide Children's Hospital
Organization: Nationwide Children's Hospital (Other)
Other Study IDs: STUDY00000910; K99NR019115-01A1 (NIH)
Record Dates: First submitted 2021-07-15; First posted 2021-07-26 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Stem Cell Transplantation
Keywords: adherence, mHealth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Primary Caregivers: Primary caregivers of children receiving Tacrolimus or cyclosporine immunosuppression for an allogeneic transplant will be introduced to the mHealth adherence app and allowed the opportunity to interact with the app alongside research staff. Following this session primary caregivers are asked to use the app at home until Day 100 or weaning of immunosuppressant, whichever is first.
  Interventions: Behavioral: mHealth adherence app

INTERVENTIONS:
Behavioral: mHealth adherence app — The mHealth app is designed to remind caregivers to give medication in the outpatient setting, track adherence, and capture real time barriers to adherence if medication is missed.

SUMMARY:
Through a mixed methods, quasi-experimental design, the study will first focus on developing a mobile health (mHealth) adherence application and evaluating usability and acceptability of the app among caregivers of children in the acute phase post-HSCT. The purpose of this project is to explore the feasibility and acceptability of a mHealth application through user testing and thematic content analysis.

ELIGIBILITY:
Inclusion Criteria:

* English-speaking
* >18 years of age

Exclusion Criteria:

* Caregivers with developmental delays or conditions that make processing and responding to verbal questions challenging/frustrating either online or in a group forum

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Primary caregivers and health care providers of children discharged during the acute phase (first 100 days) post-hematopoietic stem cell transplant (HSCT).
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2021-09-15 (Actual); Primary Completion 2023-01-31 (Actual); Study Completion 2023-01-31 (Actual)

PRIMARY OUTCOMES:
System Usability Scale (SUS) | Baseline to day 100
  The SUS is a 10-item questionnaire used to evaluate the functionality and acceptability of mHealth apps. Items are rated on a 5 point scale and final scores on the measure range from 0 to 100. Higher scores represent better functionality and acceptability. Scores of > 68 are considered above average.

CONTACTS AND LOCATIONS:
Overall Officials: Micah Skeens, PhD APRN CPNP, Principal Investigator — Abigail Wexner Research Institute at Nationwide Children's Hospital
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Skeens M, Sezgin E, Stevens J, Landier W, Pai A, Gerhardt C. An mHealth App to Promote Adherence to Immunosuppressant Medication and Track Symptoms in Children After Hematopoietic Stem Cell Transplant: Protocol for a Mixed Methods Usability Study. JMIR Res Protoc. 2022 Jul 21;11(7):e39098. doi: 10.2196/39098. PMID 35862184